CLINICAL TRIAL: NCT03863561
Title: The Skills, Confidence & Preparedness Index (SCPI) Version 3.0: An Online Version of the SCPI to Evaluate Self-Efficacy of Diabetes Management
Brief Title: The Skills, Confidence & Preparedness Index (SCPI)
Acronym: SCPI
Status: Completed | Type: Observational
Sponsor: LMC Diabetes & Endocrinology Ltd. (Other)
Responsible Party: Sponsor
Other Study IDs: SCPI
Record Dates: First submitted 2019-02-22; First posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Diabetes Mellitus
Keywords: self-management; questionnaire; diabetes education
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Waiting room sample: Patients with type 1 or type 2 diabetes attending an LMC Diabetes & Endocrinology specialist clinic in Ontario completed the SCPI in the waiting room while attending their usual appointment with their healthcare provider.
- DSME Intervention: Patients with poor glycemic control (A1C >8.0%) were enrolled into a diabetes self-management education (DSME) program. The SCPI was completed at their first and last visit and and their individual results were incorporated into the care paths that were then customized for that participant. The patient met with a diabetes educator five to seven times over the course of three to four months.
  Interventions: Behavioral: Diabetes self-management education (DSME) program

INTERVENTIONS:
Behavioral: Diabetes self-management education (DSME) program — Diabetes educators customized care paths for their patients based on their individual responses to the SCPI questions. Patients met with an educator five to seven times over the course of three to four months.
  Other Names: DSME
  Groups: DSME Intervention

SUMMARY:
The LMC Skills, Confidence and Preparedness Index (SCPI) is a tool that was developed by diabetes specialists to individualize the education/support that a healthcare provider delivers to patients with diabetes. It has been shown to have high reliability, validity and generalizability. This study assessed the validity and reliability of a revised, final version of the SCPI in a large sample of patients with type 1 and type 2 diabetes, as well as the clinical responsiveness of the SCPI to a diabetes self-management education intervention in a smaller cohort of patients with poor glycemic control.

DETAILED DESCRIPTION:
Canadian experts in diabetes care developed the Skills, Confidence & Preparedness Index (SCPI) to assess diabetes self-management in patients. The SCPI is web-based, gives immediate feedback to the healthcare provider, and is associated with glycemia. The SCPI was designed to allow a healthcare provider to individualize the education/support by assessing the three critical dimensions of self-management: knowledge of a skill; confidence in ability to change a behavior; and preparedness to begin implementing the behavior change. Two previous validation studies showed that the SCPI has high internal consistency, reliability, generalizability, and external validity.

Following further focus groups with healthcare providers and patients, the SCPI questions and response scale were edited to further optimize clarity. This study assessed the validity and reliability of a revised, final version of the LMC SCPI in a large sample of diabetes patients, as well as clinical responsiveness of the SCPI to a diabetes self-management education (DSME) program intervention.

This study recruited type 1 and type 2 patients from the waiting rooms of seven LMC Diabetes & Endocrinology specialist clinics in Ontario, Canada. Patients completed the SCPI electronically and their demographic and health information was retrieved from their electronic medical records. A smaller cohort of patients with uncontrolled glycemia were enrolled into a DSME program. Participants completed the SCPI at their baseline visit and their individual results were incorporated into the care paths that were then customized for that participant. The DSME program provided five to seven visits with a diabetes educator over three to four months. Patients completed the SCPI again at their final visit.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 1 or type 2 diabetes
* Age ≥ 18 years
* Ability to read English
* Duration of diabetes ≥ 6 months (DSME cohort only)
* A1C ≥ 8.0% (DSME cohort only)

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Waiting room cohort: adult patients with type 1 or type 2 diabetes attending their usual visit with their LMC healthcare provider
  DSME cohort: patients with type 1 or type 2 diabetes with a recent A1C ≥ 8.0%
Sampling Method: Non-Probability Sample
Enrollment: 486 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2018-12-03 (Actual); Study Completion 2018-12-03 (Actual)

PRIMARY OUTCOMES:
Internal consistency of the SCPI (Skills, Confidence & Preparedness Index) | 24-hours
  Cronbach's alpha score for the total SCPI score (minimum score 1, maximum score 7) and the three subscales (minimum score 1, maximum score 7) in the waiting room sample. A higher score indicates greater diabetes self-management.
Validity of the SCPI with HbA1c | 24-hours
  Correlation between the total SCPI score (minimum score 1, maximum score 7) and the three subscale scores (minimum score 1, maximum score 7) with HbA1c in the waiting room sample.
  A higher SCPI score indicates greater diabetes self-management.

SECONDARY OUTCOMES:
Validity of the SCPI with demographic and diabetes variables | 24-hours
  Correlation between the total SCPI score (minimum score 1, maximum score 7) and age, gender, education, ethnicity, duration of diabetes and diabetes therapy in the waiting room sample.
  A higher SCPI score indicates greater diabetes self-management.
Test-retest reliability | one week
  Applicable to patients from the waiting room sample who completed the SCPI in the clinic and again one week later. Correlation between the first total SCPI score (minimum score 1, maximum score 7) and the second total SCPI scores.
Floor/ceiling effect of the total SCPI score | 24-hours
  Assessment of a floor effect (>15% of patients with a minimum score of 1) or a ceiling effect (>15% of patients with a maximum score of 7)
SCPI completion time | 24-hours
  Mean number of minutes it took for patients to complete the SCPI
Change in SCPI score | 3 to 4 months
  Mean change in SCPI total score between the baseline visit and follow-up visit in the DSME cohort
Change in HbA1c | 3 to 4 months
  Mean change in HbA1c between the baseline visit and the follow-up visit in the DSME cohort
Association between total SCPI score and HbA1c | Baseline
  Correlation between SCPI score at baseline and HbA1c at baseline in the DSME cohort
Responsiveness of the total SCPI score to an intervention | 3 to 4 months
  Correlation between change in SCPI score and change in HbA1c in the DSME cohort

CONTACTS AND LOCATIONS:
Overall Officials: Ronnie Aronson, MD, FRCPC, FACE, Principal Investigator — LMC Diabetes & Endocrinology
Locations (7):
- Canada (7):
  - LMC Barrie, Barrie, Ontario
  - LMC Brampton, Brampton, Ontario
  - LMC Etobicoke, Etobicoke, Ontario
  - LMC Oakville, Oakville, Ontario
  - LMC Thornhill, Thornhill, Ontario
  - LMC Scarborough, Toronto, Ontario
  - LMC Bayview, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mbuagbaw L, Aronson R, Walker A, Brown RE, Orzech N. The LMC Skills, Confidence & Preparedness Index (SCPI): development and evaluation of a novel tool for assessing self-management in patients with diabetes. Health Qual Life Outcomes. 2017 Jan 31;15(1):27. doi: 10.1186/s12955-017-0606-z. PMID 28143548
- [Background] Aronson R, Brown RE, Jiandani D, Walker A, Orzech N, Mbuagbaw L. Assessment of self-management in patients with diabetes using the novel LMC Skills, Confidence and Preparedness Index (SCPI). Diabetes Res Clin Pract. 2018 Mar;137:128-136. doi: 10.1016/j.diabres.2017.10.028. Epub 2017 Oct 31. PMID 29097289
- [Background] Aronson R, Orzech N, Ye C, Brown RE, Goldenberg R, Brown V. Specialist-Led Diabetes Registries and Prevalence of Poor Glycemic Control in Type 2 Diabetes: The Diabetes Registry Outcomes Project for A1C Reduction (DROP A1C). Diabetes Care. 2016 Oct;39(10):1711-7. doi: 10.2337/dc15-2666. Epub 2016 Aug 11. PMID 27515966
- [Background] Aronson R, Orzech N, Ye C, Goldenberg R, Brown V. Specialist-led diabetes registries and predictors of poor glycemic control in type 2 diabetes: Insights into the functionally refractory patient from the LMC Diabetes Registry database. J Diabetes. 2016 Jan;8(1):76-85. doi: 10.1111/1753-0407.12257. Epub 2015 Mar 24. PMID 25565383
- [Derived] Aronson R, Li A, Brown RE, Walker A, Lyons A, Orzech N. Optimizing Diabetes Self-management Using the Novel Skills, Confidence, and Preparedness Index (SCPI). Diabetes Care. 2019 Oct;42(10):1873-1878. doi: 10.2337/dc19-0699. Epub 2019 Aug 9. PMID 31399439